CLINICAL TRIAL: NCT01683513
Title: Prospective Randomized Trial on GnRH Agonist Triggering Versus hCG Triggering in IVF Stimulation in PCOS Patients
Brief Title: Trial Comparing hCG Triggering Versus GnRH Agonist Triggering in PCOS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Jan Palfijn Gent (Other)
Collaborators: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Dr. Decleer Wim, gynecologist, AZ Jan Palfijn Gent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr. Decleer W
Record Dates: First submitted 2012-08-23; First posted 2012-09-12 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Infertility; PCOS
Keywords: OHSS; mataphase II oocytes (MII); good quality embryo's; pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- humaan chorion gonadotropine (No Intervention): ovulation induction with 5000E hCG
- GnRH agonist + 1500E hCG (Active Comparator): ovulation induction with GnRH agonist and 1500E hCG one hour after egg retrieval
  Interventions: Drug: GnRh agonist +1500E hCG

INTERVENTIONS:
Drug: GnRh agonist +1500E hCG — ovulation induction with GnRh agonist and 1500E hCG one hour after egg retrieval
  Arms: GnRH agonist + 1500E hCG

SUMMARY:
In this study the investigators compare the traditional way of triggering with a new way in patients with Poly Cystic Ovary Syndrome (PCOS). This to reduce the risque of Ovary Hyper Stimulation Syndrome (OHSS) in In Vitro Fertilization/ IntraCytoplastic Sperm Injection (IVF/ ICSI) treatment. The investigators also compare the number of mature oocytes, embryo's and pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* ICSI patients below 38 years
* 1, 2 and 3e IVF cycle
* Body Mass Index (BMI) less than 32
* PCOS patients

Exclusion Criteria:

* endocrinal diseases or problems

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
MII oocytes | patients will be followed during the stimulation with an average of 10 days
  The number of mature oocytes retrieved after stimulation without creating OHSS
2 Pro Nuclei (2PN) fertilization | 24h after ICSI
  laboratory follow up of the fertilized egg during the first 24h

SECONDARY OUTCOMES:
implantation rate | 12 weeks
  The number of pregnancies obtained wich still is the most important issue for the patients
OHSS | one month with oocyte retrieval in the middle
  patient follow up according to subjective complaints and objective measures

CONTACTS AND LOCATIONS:
Overall Officials: Wim Decleer, gynecologist, Principal Investigator — IVF Centrum Jan Palfijn Gent
Locations (1):
- AZ Jan Palfijn, Ghent, Oost-vlaanderen, Belgium